CLINICAL TRIAL: NCT05561400
Title: Combining Cerebellar tDCS and Constraint-induced Language Therapy in Non-fluent Aphasia: a Novel Approach to Target Discourse
Brief Title: Combining tDCS and CILT in Non-fluent Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SLP-2022-29906
Record Dates: First submitted 2022-06-23; First posted 2022-09-30 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Aphasia; Non-fluent Aphasia; Stroke; Brain Injuries
Keywords: transcranial direct current stimulation (tDCS); non-invasive brain stimulation (NIBS); aphasia; constraint-induced language therapy (CILT)
MeSH Terms: conditions — Aphasia; Aphasia, Broca; Stroke; Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Sham controlled blinded crossover design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Real tDCS (Active Comparator): the participant receives real tDCS to the right cerebellum during behavioral intervention (CILT)
  Interventions: Device: tDCS
- Sham tDCS (Placebo Comparator): the participant receives sham tDCS to the right cerebellum during behavioral intervention (CILT)
  Interventions: Other: Placebo

INTERVENTIONS:
Device: tDCS — 5x5 saline-soaked sponge electrodes will be used with the cathode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the anode will be placed on the right shoulder. The electrode placement will be the same across both conditions.
  Arms: Real tDCS
Other: Placebo — sham tDCS to the right cerebellum
  Arms: Sham tDCS

SUMMARY:
The long-term goal of this work is to determine if combining a highly intensive, task-specific behavioral language intervention with modulation of the efferent cerebellar-cortical pathway using transcranial direct current stimulation (tDCS) has a positive influence on discourse, verbal fluency and working memory in individuals with non-fluent aphasia after stroke. And if these changes can be related to neuroplastic change in the cerebellar cortical pathway indirectly measured through neurophysiologic changes using spectral electroencephalogram (EEG). The initial phase includes the proposed pilot study data from which will be used to inform a larger clinical trial. The primary aims of this pilot are to 1) determine the effect of combining cerebellar tDCS with constraint-induced language therapy (CILT) on language as measured by a verbal fluency task and discourse task in a small population and 2) identify the tolerance of the intervention and barriers to participation measured by the adverse events questionnaire that will inform the methodology of a larger study. The secondary aims include estimating the size of the treatment effect on 1) delta percentage in F3, F7 and Fp1 compared to F4, F8, and Fp2 using resting state EEG spectral analysis and coherence, 2) working memory as measured by the score on the n-back test and 3) quality of life as measured by the Stroke Aphasia Quality of Life survey tool. The secondary aims will be used to determine the utility of these measures in a larger clinical trial.

This is a prospective, crossover study, sham-controlled intervention study with two intervention conditions delivered across 6 intervention sessions (3x/week for two weeks) with a 4-week washout in between. Conditions include: 1) sham cerebellar tDCS and 2) real cerebellar tDCS delivered at 2mA across 20 minutes. Each of these will be delivered during CILT intervention with a licensed, certified speech-language pathologist trained in CILT. Once tDCS stimulation has ended, CILT will continue to be delivered for an additional 25 minutes. Assessments of discourse, verbal fluency, working memory and EEG spectral analysis will be conducted at four timepoints, before and after each intervention phase.

DETAILED DESCRIPTION:
This is a prospective sham-controlled, cross-over design. Eligible participants must be over the age of 18 years, be > least 6 months post unilateral cortical stroke and diagnosed with mild to moderate non-fluent aphasia. Additional inclusion/exclusionary criteria have been specified in and approved by the IRB. Six to seven participants are expected to be recruited and screened, with the goal to enroll and complete the study with four individuals who will be randomly assigned to receive either sham or real condition first. The two intervention conditions include: 1) andodal tDCS (2mA) to the right posterior-lateral cerebellum and 2) sham tDCS to the right posterior-lateral cerebellum. The participants will receive 20 minutes of tDCS (sham or real) during CILT followed by an additional 25 minutes of CILT alone. Each condition will be administered 3 days per week for two weeks for a total of 6 intervention sessions with a 4-week washout period between.

For tDCS (TCT-Research Version tDCS Stimulator, Hong Kong), two 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting the posterior lateral cerebellum and the cathode will be placed on the right shoulder. The electrode placement will be the same across both conditions. The CILT behavioral intervention will be led by a certified, licensed speech-language pathologist and a graduate student researcher and will follow the guidelines of CILT.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years
* history of stroke
* diagnosed with non-fluent aphasia.
* be able to independently understand simple directions,
* use some speech to communicate,
* have access to reliable transportation (including taxi and/or other transportation services),
* fluent in English.

Exclusion Criteria:

* Pregnancy,
* history of seizures,
* any metal implants in the body (excluding dental fillings),
* history of migraines,
* psoriasis or eczema affecting the scalp,
* history of a head injury such as a concussion
* diagnosis of a mental health or neurological condition/disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharyl A Samargia-Grivette, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Duluth, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Real tDCS First: The participant receives the real tDCS condition and then crosses over to the sham condition.
  Real tDCS condition: paricipant received real tDCS to the right cerebellum at 2mA for 20 minutes during behavioral intervention (CILT)
  tDCS: 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at 2mA for 20 minutes.
- Sham tDCS First: The participant receives the sham tDCS condition first and then crosses over to the real tDCS condition.
  Sham tDCS: participant receives sham/placebo stimulation to the right cerebellum during behavioral intervention (CILT)
  Participant is still fit wth 5x5cm saline soaked electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at "sham" condition which ramps up for ~60 seconds of stimulation before ramping down.
Period: Overall Study
Arm/Group | Real tDCS First | Sham tDCS First
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS First | Sham tDCS First | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8) | 61 (5.65) | 61.6 (6.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Discourse: Picture Description
Description: Picture Description using Main Concept Analysis (MCA), a reliable, valid method of discourse analysis. It captures a participant's ability to state the main points/highlights of a sequential story. Responses to the "Broken Window" picture sequence, a normed and standardized task are recorded as accurate and complete (3 points), accurate and incomplete (2 points), inaccurate and complete (2 points), inaccurate and incomplete (1 point) or absent (0points). The minimum score is 0 and the maximum score is 24. There are no subscales. The higher the score, the better the performance. Scores reported for individual participants are raw scores.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: occurred at Visit 2 (after consent)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Real tDCS Condition First: The participant receives the real tDCS condition and then crosses over to the sham condition.
  Real tDCS condition: paricipant received real tDCS to the right cerebellum at 2mA for 20 minutes during behavioral intervention (CILT)
  tDCS: 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at 2mA for 20 minutes.
- Sham tDCS Condition First: The participant receives the sham tDCS condition and then crosses over to the real condition.
  Sham condition: paricipant received sham tDCS to the right cerebellum at 2mA for 20 minutes during behavioral intervention (CILT)
  Sham tDCS: 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at 2mA for 20 minutes. tDCS set at "sham" mode Sham is the placebo
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 10 (2.82) | 5.66 (2.08)

2. Primary Outcome: Discourse Analysis: Picture Description
Description: as for outcome 1
Time Frame: Follow up 1: Visit 9. 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: Raw Score/Points
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
Raw Score/Points | 7.66 (8.02) | 13 (1.41)

3. Primary Outcome: Discourse: Picture Description
Description: Picture Description using Main Concept Analysis (MCA), a reliable, valid method of discourse analysis. It captures a participant's ability to state the main points/highlights of a sequential story. Responses to the "Broken Window" picture sequence, a normed and standardized task are recorded as accurate and complete (3 points), accurate and incomplete (2 points), inaccurate and complete (2 points), inaccurate and incomplete (1 point) or absent (0points). The minimum score is 0 and the maximum score is 24. There are no subscales. The higher the score, the better the performance. Scores reported for individual participants are raw scores.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after Follow up 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 7 (6.08) | 14 (8.48)

4. Primary Outcome: Discourse Analysis: Picture Description
Description: as for outcome 3
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1 and 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 11.66 (10.40) | 10 (2.82)

5. Primary Outcome: Discourse Analysis: Story Retell
Description: Story Retell using Main Concept Analysis (MCA), counts of the number of main ideas or propositions that are necessary for successful discourse. Responses to the "Cinderella" story retell task, a normed and standardized task will be recorded using the standardized "counts" or "raw score" main concept analysis scoring system. The minimum score is 0 and the maximum score is 102. There are no subscales for this measure. Responses are scored using the following rubric: accurate and complete (3 points), accurate and incomplete (2 point), inaccurate and complete (2 point) inaccurate and incomplete (1 points) or absent (0 points). The higher the score, the better the performance. Participant scores are reported as raw scores.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: occurred at Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 31 (29.61) | 23 (7.07)

6. Primary Outcome: Discourse Analysis: Story Retell
Description: as for outcome 5
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 31.66 (29.73) | 31 (25.45)

7. Primary Outcome: Discourse Analysis: Story Retell
Description: Story Retell using Main Concept Analysis (MCA), counts of the number of main ideas or propositions that are necessary for successful discourse. Responses to the "Cinderella" story retell task, a normed and standardized task will be recorded using the standardized "counts" or "raw score" main concept analysis scoring system. The minimum score is 0 and the maximum score is 102. There are no subscales for this measure. Responses are scored using the following rubric: accurate and complete (3 points), accurate and incomplete (2 point), inaccurate and complete (2 point) inaccurate and incomplete (1 points) or absent (0 points). The higher the score, the better the performance. Participant scores are reported as raw scores.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after follow up 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 33.66 (30.66) | 28.5 (14.84)

8. Primary Outcome: Discourse Analysis: Story Retell
Description: as for outcome 7
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1 and 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 35 (30.41) | 26 (16.97)

9. Primary Outcome: Discourse Analysis: Procedural
Description: Procedural Discourse using Main Concept Analysis (MCA), counts of the number of main ideas or propositions that are necessary for successful procedural discourse. Responses "how to make a peanut butter sandwich" task, a normed and standardized task will be recorded using the standardized "counts" or "raw score" main concept analysis scoring system. The minimum score is 0 and the maximum score is 30. There are no subscales. The higher the score, the better the performance. Participant responses are scored using a rubric: accurate and complete (3 points), accurate and incomplete (2 point)s, inaccurate and complete (2 points), inaccurate and incomplete (1 point) or absent (0 points). Participant scores are reported as raw scores. There are no subscales for this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: Visit 2
Measure: Mean (Standard Deviation); unit: Raw Score/Points
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
Raw Score/Points | 10 (9.53) | 17 (7.07)

10. Primary Outcome: Discourse Analysis: Procedural
Description: as for outcome 9
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 11.66 (10.40) | 14 (0)

11. Primary Outcome: Discourse Analysis: Procedural
Description: Procedural Discourse using Main Concept Analysis (MCA), counts of the number of main ideas or propositions that are necessary for successful procedural discourse. Responses "how to make a peanut butter sandwich" task, a normed and standardized task will be recorded using the standardized "counts" or "raw score" main concept analysis scoring system. The minimum score is 0 and the maximum score is 30. There are no subscales. The higher the score, the better the performance. Participant responses are scored using a rubric: accurate and complete (3 points), accurate and incomplete (2 point)s, inaccurate and complete (2 points), inaccurate and incomplete (1 point) or absent (0 points). Participant scores are reported as raw scores. There are no subscales for this measure.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after follow up 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 14.33 (9.29) | 15 (2.82)

12. Primary Outcome: Discourse Analysis: Procedural
Description: as for outcome 11
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1 and 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 11.66 (10.11) | 14.5 (3.53)

13. Primary Outcome: Verbal Fluency: Semantic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many animals as they can in one minute. Norms for healthy adults is between 18-20 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17 items. The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: Visit 2
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 12.33 (12.01) | 18.5 (2.12)

14. Primary Outcome: Verbal Fluency: Semantic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many animals as they can in one minute. Norms for healthy adults is between 18-20 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17 items.The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 15.33 (13.31) | 17.5 (6.36)

15. Primary Outcome: Verbal Fluency: Semantic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many animals as they can in one minute. Norms for healthy adults is between 18-20 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17 items.The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after Follow up 1
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 10.66 (11.01) | 16 (9.89)

16. Primary Outcome: Verbal Fluency: Semantic
Description: as for outcome 15
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1, 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 12 (10.81) | 16 (12.72)

17. Primary Outcome: Verbal Fluency: Phonemic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many words they can that start with either /f/ in one minute. Norms for healthy adults is between 25-35 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17. The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: Visit 2
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 4.66 (2.51) | 8.5 (4.94)

18. Primary Outcome: Verbal Fluency: Phonemic
Description: as for outcome 17
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 4 (3.6) | 14.5 (9.19)

19. Primary Outcome: Verbal Fluency: Phonemic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many words they can that start with either /f/ in one minute. Norms for healthy adults is between 25-35 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17.The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after Follow up 1
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 3 (2.64) | 12.5 (13.43)

20. Primary Outcome: Verbal Fluency: Phonemic
Description: Verbal Fluency is a normed and standardized task of working memory and word recall. Participant will name as many words they can that start with either /f/ in one minute. Norms for healthy adults is between 25-35 items listed within the one minute timeframe. The number of items listed is the participants raw score. The higher the score, the better the performance. A score considered "no concerns" is >17. The minimum score is 0. There is no maximum score as this is a timed measure. There is no subscales for this measure.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1 and 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: raw score number of items named
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
raw score number of items named | 4 (4) | 18.5 (13.43)

21. Secondary Outcome: Working Memory
Description: To measure working memory, the participant will complete the 2 n-back test. The score represents the raw score which is calculated as the total possible minus errors, which is called the accuracy score. The higher the score the better. In healthy adults, the average accuracy score is between 50%-75%. A minium accuracy score is 0 and the maximum score is 100%. There are no subscales in this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: Visit 2
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
percentage of accuracy | 55.33 (20.52) | 70 (18.34)

22. Secondary Outcome: Working Memory
Description: To measure working memory, the participant will complete the 2 n-back test. The score represents the raw score which is calculated as the total possible minus errors, which is called the accuracy score. The higher the score the better. In healthy adults, the average accuracy score is between 50%-75%.A minium accuracy score is 0 and the maximum score is 100%. There are no subscales in this measure.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
percentage of accuracy | 81.66 (16.07) | 71.5 (40.30)

23. Secondary Outcome: Working Memory
Description: To measure working memory, the participant will complete the 2 n-back test. The score represents the raw score which is calculated as the total possible minus errors, which is called the accuracy score. The higher the score the better. In healthy adults, the average accuracy score is between 50%-75%. A minium accuracy score is 0 and the maximum score is 100%. There are no subscales in this measure.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after Follow up 1
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
percentage of accuracy | 74.33 (22.89) | 76.5 (2.12)

24. Secondary Outcome: Working Memory
Description: as for outcome 23
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1 and 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: percentage of accuracy
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
percentage of accuracy | 77.33 (11.84) | 75 (35.35)

25. Secondary Outcome: Stroke Aphasia Quality of Life (SA-QOL)
Description: Stroke Aphasia Quality of Life (SA-QOL) is a participant perception survey. Response scale between 1 and 5. 1=Total help / couldn't do it at all / strongly agree, 2=a lot of help / a lot of trouble / moderately agree, 3= some help / some trouble / neight agree nor disagree, 4= a little help / a little trouble / moderately disagree or 5= no help needed / no trouble at all / strongly disagree. 3 subscales:
  Physical, the total number of questions is 16, minimum score is 16 and the maximum score is 80.
  Communication, the total number of qustions is 7, minimum score is 7 and maximum score is 35 Psychosocial, the total number of questions is 16, minimum score is 16 and maximum score is 80 Scores from these subscales are totalled and divided by 39 to get the score. Total minimum score is 1 and total maximum score is 5 Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Baseline 1: Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 3.74 (0.313) | 3.37 (1.10)

26. Secondary Outcome: Stroke Aphasia Quality of Life (SA-QOL)
Description: Stroke Aphasia Quality of Life (SA-QOL) is a participant perception survey. Scale is between 1 and 5. 1=Total help / couldn't do it at all / strongly agree, 2=a lot of help / a lot of trouble / moderately agree, 3= some help / some trouble / neight agree nor disagree, 4= a little help / a little trouble / moderately disagree or 5= no help needed / no trouble at all / strongly disagree. 3 subscales:
  Physical, total number of questions is 16, minimum score is 16 and the maximum score is 80.
  Communication, total number of qustions is 7, minimum score is 7 and maximum score is 35 Psychosocial, the total number of questions is 16, minimum score is 16 and maximum score is 80 Scores from these subscales are totalled and divided by 39 to get the score. Total minimum score is 1 and total maximum score is 5. The higher the score reflect better quality of life.
  Baseline 1 and Follow up 1 refer to the first intervention condition in the cross over sequence.
Time Frame: Follow up 1: Visit 9: 2 weeks after Baseline 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 3.74 (0.27) | 3.77 (0.65)

27. Secondary Outcome: Stroke Aphasia Quality of Life (SA-QOL)
Description: Stroke Aphasia Quality of Life (SA-QOL) is a participant perception survey. Response scale is between 1 and 5. 1=Total help / couldn't do it at all / strongly agree, 2=a lot of help / a lot of trouble / moderately agree, 3= some help / some trouble / neight agree nor disagree, 4= a little help / a little trouble / moderately disagree or 5= no help needed / no trouble at all / strongly disagree. There are 3 subscales:
  Physical, total number of questions is 16, minimum score is 16 and the maximum score is 80.
  Communication, the total number of qustions is 7, minimum score is 7 and maximum score is 35 Psychosocial, the total number of questions is 16, minimum score is 16 and maximum score is 80 Scores from these subscales are totalled and divided by 39 to get the score. Total minimum score is 1 and total maximum score is 5. The higher the score reflect better quality of life.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Baseline 2: Visit 10. 6 weeks after Baseline 1 and 4 weeks after Follow up 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 4.00 (0.69) | 3.81 (0.707)

28. Secondary Outcome: Stroke Aphasia Quality of Life (SA-QOL)
Description: Stroke Aphasia Quality of Life (SA-QOL) is a participant perception survey. Response scale is between 1 and 5. 1=Total help / couldn't do it at all / strongly agree, 2=a lot of help / a lot of trouble / moderately agree, 3= some help / some trouble / neight agree nor disagree, 4= a little help / a little trouble / moderately disagree or 5= no help needed / no trouble at all / strongly disagree. There are 3 subscales:
  Physical, the total number of questions is 16, minimum score is 16 and the maximum score is 80.
  Communication, the total number of qustions is 7, minimum score is 7 and maximum score is 35 Psychosocial, the total number of questions is 16, minimum score is 16 and maximum score is 80 Scores from these subscales are totalled and divided by 39 to get the score. Total minimum score is 1 and total maximum score is 5. The higher the score reflect better quality of life.
  Baseline 2 and Follow up 2 reflect the second intervention in the cross over sequence.
Time Frame: Follow up 2: Visit 17. 8 weeks after Baseline 1, 6 weeks after Follow up 1, 2 weeks after Baseline 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Real tDCS Condition First | Sham tDCS Condition First
Number analyzed (Participants) | 3 | 2
score on a scale | 4.15 (0.64) | 3.75 (0.94)

ADVERSE EVENTS:
Time Frame: Each participant was asked to report adverse events from the following list: headache, neck pain, scalp pain, tingling, itching, burning sensation, skin redness, sleepiness, lack of concentration, change of mood following all intervention sessions. Each participant was seen for a total of 12 intervention sessions (6 using real tDCS and 6 using sham tDCS). Each participant was asked to report adverse effects immediately following each intervention session.
Description: The standard adverse events reported when using tDCS include: headache, neck pain, scalp pain, tigling, itching, burning sensation, skin redness, sleepiness, lack of concentration, change of mood. Adverse events were reported following each intervention session (12 in total). Partcipants were monitored for adverse effects through the course of the study (2 weeks during one condition and then 2 weeks during the second condition). Adverse events monitoring was not done during the wash out period.
Groups:
- Real tDCS Condition: Real tDCS condition: paricipant received real tDCS to the right cerebellum at 2mA for 20 minutes during behavioral intervention (CILT)
  tDCS: 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at 2mA for 20 minutes.
- Sham tDCS Condition: Sham condition: paricipant received sham tDCS to the right cerebellum at 2mA for 20 minutes during behavioral intervention (CILT)
  Sham tDCS: 5x5 saline-soaked sponge electrodes will be used with the anode placed over the right cerebellar hemisphere; 1cm under and 4cm lateral of the inion targeting lobule VII and the cathode placed on the right deltoid. tDCS was set at 2mA for 20 minutes. tDCS set at "sham" mode Sham is the placebo
Arm/Group | Real tDCS Condition | Sham tDCS Condition
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real tDCS Condition (N=5) | Sham tDCS Condition (N=5)
Headache (General disorders) | 1 (3) | 1 (6)
Neck Pain (General disorders) | 0 (0) | 1 (1)
Tingling sensation (General disorders) | 3 (10) | 0 (0)
Itching (General disorders) | 2 (3) | 0 (0)
Burning sensation (General disorders) | 1 (1) | 0 (0)
skin redness (General disorders) | 1 (6) | 1 (1)
sleepiness (General disorders) | 2 (3) | 1 (2)
Trouble concentrating (General disorders) | 2 (5) | 2 (4)
acute change of mood (General disorders) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT05561400/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05561400/ICF_001.pdf